CLINICAL TRIAL: NCT02548923
Title: Dexmedetomidine Versus Propofol for Prolonged Sedation in Critically Ill Trauma and Surgical Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Responsible Party: Principal Investigator, Brian Daley, Professor, University of Tennessee Graduate School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UTMCKTRAUMA1
Record Dates: First submitted 2015-08-14; First posted 2015-09-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine group (Active Comparator): Patients who received dexmedetomidine for sedation
  Interventions: Drug: Dexmedetomidine
- propofol group (No Intervention): Patients who received propofol for sedation

INTERVENTIONS:
Drug: Dexmedetomidine — comparison to propofol
  Other Names: Propofol
  Arms: dexmedetomidine group

SUMMARY:
The purpose of this study is to assess the efficacy of dexmedetomidine versus propofol for prolonged sedation in trauma and surgical patients.

DETAILED DESCRIPTION:
Design: Open-label, single-center prospective study. Setting: Trauma/Surgical Intensive Care Unit (TSICU) at a Level I academic trauma center.

Patients: Patients 18 years of age or older requiring mechanical ventilation and admitted to the TSICU Interventions: Patients were randomly assigned based on unit bed location to receive dexmedetomidine or propofol for sedation.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included in the study if they were 18 years of age or older,
* mechanically ventilated,
* placed on the institutional sedation protocol,
* expected to require sedation lasting 24 hours after randomization, and
* admitted to the TSICU and followed by the Trauma/Surgical Service.

Exclusion Criteria:

Patients were excluded for any of the following:

* 72 hours or greater since sedation protocol initiation,
* treatment per the institutional traumatic brain injury (TBI) protocol,
* concomitant continuous infusion of a neuromuscular blocking agent,
* heart rate less than 50 beats per minute,
* mean arterial pressure less than 55 mmHg despite fluid resuscitation and vasopressors, and
* use of other alpha-2 agonists within 24 hours of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Duration of Mechanical Ventilation | ICU stay
  An average of 10 days

SECONDARY OUTCOMES:
Mortality | Hospital length of stay
  An average of 21 days
proportion of time in target sedation | ICU length of stay
  AN average of 10 days
incidence of delirium | ICU length of stay
  An average of 10 days
hypotension | ICU length of stay
bradycardia | ICU length of stay
  AN Average of 10 days
ICU and hospital length of stay | hospital length of stay
  An average of 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Medical Center, Knoxville, Tennessee, United States